CLINICAL TRIAL: NCT01399827
Title: Omega-3 Fatty Acid Supplementation to ADHD Pharmacotherapy in ADHD Adults With DESR Traits: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial
Brief Title: Omega-3 Fatty Acid Supplementation to ADHD Pharmacotherapy in ADHD Adults With Deficient Emotional Self-Regulation Traits
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Scientific Coordinator of the Adult ADHD Program, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-P-002435
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Deficient Emotional Self-Regulation (DESR)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Lisdexamfetamine Dimesylate; Dextroamphetamine; Adderall; Amphetamine; Atomoxetine Hydrochloride; Dexmethylphenidate Hydrochloride; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Fatty Acids (Active Comparator): 1060 mg EPA Omega-3 Fatty Acids
  Interventions: Drug: ADHD Medication; Drug: Omega-3 Fatty Acids
- Placebo (Placebo Comparator)
  Interventions: Drug: ADHD Medication

INTERVENTIONS:
Drug: ADHD Medication — For those subjects not on stable ADHD treatment (defined as a stable, effective dose for at least one month, determined by the study clinician, of a medication that is FDA approved to treat ADHD), OROS-Methylphenidate will be openly prescribed. Subjects on a stable dose of medication for ADHD will be instructed to continue on their current dose of medication.
  Other Names: Methylphenidate extended release (OROS-MPH); Concerta; Vyvanse; Dextroamphetamine; Adderall; Mixed Amphetamine Salts; Amphetamine; Strattera; Atomoxetine; Focalin; Dexmethylphenidate
Drug: Omega-3 Fatty Acids — Omega-3 Fatty Acids prescribed to participants randomized to active medication. They may be randomized to receive 1060mg of EPA (2 capsules containing 530mg EPA and 137mg DHA). Dosage will remain constant throughout study.
  Other Names: Nordic Natural EPA Xtra
  Arms: Omega-3 Fatty Acids

SUMMARY:
The purpose of this study is to a) assess the efficacy of omega-3 fatty acids in the treatment of Deficient Emotional Self-Regulation (DESR) among stimulant treated Attention Deficit Hyperactivity Disorder (ADHD) adults, b) assess the side effect profile of omega-3 fatty acids in the treatment of DESR among stimulant treated ADHD adults, c) assess effects of omega-3 fatty acid supplementation on ADHD symptoms and associated features in stimulant treated ADHD adults, and d) predict value of fatty acids present in red blood cell membranes. This study will be a 12-week trial with adults 18-55 years of age with ADHD and symptoms of DESR.

ELIGIBILITY:
Inclusion Criteria

1. Male or female adults ages 18-55 years.
2. A diagnosis of childhood onset Attention Deficit Hyperactivity Disorder, according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) based on clinical assessment. Childhood onset will be defined according to established research criteria, requiring onset of two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12.
3. A score of 24 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS), or, for those individuals stably treated with a medication approved by the Food and Drug Administration for ADHD, a Clinical Global Impression (CGI) ADHD severity score of no greater than 4 ("moderately ill").

   Those subjects treated with traditional ADHD pharmacotherapy must be on a stable, effective dose (per clinician evaluation) of an FDA-approved treatment for ADHD for at least one month at the time of enrollment.
4. A Deficient Emotional Self Regulation (DESR) T-score on the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Emotional Control Scale of at least 65 and/or a score of 99 or more on the DESR.

Exclusion Criteria

1. For those subjects not treated for their ADHD at the time of enrollment, a history of non-response or intolerance to methylphenidate at adequate doses as determined by the clinician.
2. A history of intolerance to omega-3 fatty acids as determined by the clinician.
3. Pregnant or nursing females.
4. Serious, unstable medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinologic (thyroid), neurologic (seizure), immunologic, or hematologic disease.
5. Glaucoma.
6. Clinically unstable psychiatric conditions including suicidality, homicidality, bipolar disorder, psychosis, or lifetime history of a clinically serious condition potentially exacerbated by a stimulant such as mania, or psychosis.
7. Tics or a family history or diagnosis of Tourette's syndrome.
8. Current (within 3 months) DSM-IV criteria for abuse or dependence with any psychoactive substance other than nicotine.
9. Allergies to fish or shellfish; multiple adverse drug reactions.
10. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
11. Current use of Monoamine Oxidase (MAO) Inhibitor or use within the past two weeks.
12. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (NA) — There is no standard deviation because there was only one participant. | 21 (NA) — There is no standard deviation because there was only one participant. | 34.5 (19.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 1 | 0 | 1
  Race: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Endpoint on the BRIEF-A Emotional Control Scale
Description: The BRIEF-A is a 75-item questionnaire that assesses and adult's cognitive, emotional, and behavioral functions within the past month. The subject rates each question on a 3-point scale (1=Never, 2=Sometimes, 3=Often). Raw scores are calculated and used to generate T-scores for 8 scales (Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials), 2 summary index scales (Behavioral Regulation Index and Metacognition Index), and one scale reflecting overall functioning (Global Executive Composite). T-scores range from 30 to 100, with scores ≥65 indicating clinical impairment. A reduction in score indicates improvement.
Time Frame: Baseline to 12 weeks
Measure: Number; unit: T-Score
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 1 | 1
T-Score | -7 | -33

2. Secondary Outcome: Efficacy Measured by Mean Change From Baseline to Endpoint on Adult ADHD Investigator Rating Scale (AISRS) Total Score
Description: The Adult ADHD Investigator Rating Scale (AISRS) measures ADHD symptoms in adults. This scale is an investigator rated scale. Higher scores on this scale indicate more severe ADHD-like symptoms. Patients symptoms are rated as "never", "rarely", "sometimes", "often", or "very often" by the investigator. Total score ranges from 0 to 54. T-scores range from 30 to 100, with scores ≥65 indicating clinical impairment. A reduction in score indicates improvement.
Time Frame: baseline to 12 weeks
Measure: Number; unit: T-Score
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 1 | 1
T-Score | -14 | -23

3. Secondary Outcome: Efficacy Measured by Mean Change From Baseline to Endpoint on Clinical Global Impression (CGI) Scale
Description: The Clinical Global Impression (CGI) is a 3-item observer-rated scale that measures illness severity (CGIS), global improvement or change (CGIC) and therapeutic response (CGIE). Scores range from 0 to 7 on each subscale. Total scores range from 0 to 21. T-scores range from 30 to 100, with scores ≥65 indicating clinical impairment. A reduction in score indicates improvement.
Time Frame: baseline to 12 weeks
Measure: Number; unit: T-Score
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 1 | 1
T-Score | 5 | 1

4. Secondary Outcome: Efficacy Measured by Mean Change From Baseline to Endpoint on BRIEF-A Subscales
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Measure: Number; unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale
  Change in BRIEF-A Inhibit Scale T-Scores from Base | -14 | -28
  Change in BRIEF-A Shift Scale T-Scores from Baseli | 0 | -13
  Change in BRIEF-A Self Monitor Scale T-Scores from | 0 | -13
  Change in BRIEF-A Initiate Scale T-Scores from Bas | -17 | -9
  Change in BRIEF-A Working Memory Scale T-Scores fr | -11 | -30
  Change in BRIEF-A Plan/Organize Scale T-Scores fro | -11 | -19
  Change in BRIEF-A Task Monitor Scale T-Scores from | -5 | -32
  Change in BRIEF-A Organization of Materials Scale | -6 | -22
  Change in BRIEF-A BRI Scale T-Scores from Baseline | -7 | -29
  Change in BRIEF-A MI Scale T-Scores from Baseline | -12 | -46
  Change in BRIEF-A GEC Scale T-Scores from Baseline | -11 | -29

5. Secondary Outcome: Efficacy Measured by Mean Change From Baseline to Endpoint on the Global Assessment of Functioning (GAF) Scale
Description: The Global Assessment of Functioning (GAF) scale is used to rate how serious a mental illness may be. Lower scores on this scale indicate a lower level of functioning and higher severity of symptoms. Total scores range from 0 to 100.
Time Frame: baseline to 12 weeks
Measure: Number; unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | 11 | 8

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Omega-3 Fatty Acids | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acids (N=1) | Placebo (N=1)
Facial discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Fish Body Odor (General disorders) | 1 (3) | 0 (0)
Headaches (General disorders) | 1 (1) | 0 (0)
Personality Differences (Psychiatric disorders) | 1 (2) | 0 (0)
Eye Discomfort (Eye disorders) | 1 (3) | 0 (0)
Viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Puffiness at eye (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Low appetite (Gastrointestinal disorders) | 0 (0) | 1 (3)
Jittery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT01399827/Prot_SAP_000.pdf